CLINICAL TRIAL: NCT05658653
Title: Measuring the Clinical Utility of Aegis's Chronic Disease Management Test Among VillageMD Providers: A CPV Randomized Control Trial
Brief Title: Clinical Utility of CDMT Among VillageMD Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00064387
Record Dates: First submitted 2022-12-02; First posted 2022-12-21 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Chronic Disease; Drug Drug Interaction; Medication Adherence
MeSH Terms: conditions — Chronic Disease; Medication Adherence

STUDY DESIGN:
Intervention Model Description: The study will enroll physicians and care providers practicing in the VillageMD health system. Participants are randomly assigned to either control or intervention 1 arms upon enrollment. All eligible and consented participants will complete two rounds of three patient simulations.
  The intervention arm only will receive educational material about the CDMT test in between these two rounds. Intervention arm participants only will receive the CDMT test results whether they select it or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Practice (No Intervention): The Control group treats their simulated patients using standard practice and has no introduction to the new CDMT test.
- Chronic Disease Management Test (CDMT) (Experimental): The intervention will receive information regarding the CDMT test and will be given the test results, whether selected or not, in Round 2 of CPV administration.
  Interventions: Other: Educational Materials for Chronic Disease Management Test (CDMT)

INTERVENTIONS:
Other: Educational Materials for Chronic Disease Management Test (CDMT) — These materials detail what the test does, how it is used, the validity and specifications of the test, and how to read its test report.
  Arms: Chronic Disease Management Test (CDMT)

SUMMARY:
This is a health system-level research study of physicians and care providers. The purpose of this study is to assess the clinical evaluation and management (drug, procedures, counseling, and other) of a subset of common patient care indications.

DETAILED DESCRIPTION:
The results of this study could contribute to improved quality of care for patients by encouraging better care practices and adherence to evidence-based guidelines. The data from this study will be submitted to a national journal for publication. The study plans to enroll up to 150 physicians.

Upon consenting and agreeing to participate in this study, participants will be asked to care for 3 simulated patient cases, known as Clinical Performance and Value Vignettes (CPV®). CPVs describe patients physicians typically encounter in their daily practice and are not meant to be difficult. In each vignette, physicians are asked to share their expected care through 5 domains: 1) history, 2) physical exam, 3) diagnostic workup, 4) diagnosis, and 5) treatment and follow-up. Each case takes approximately 15-20 minutes to complete and the investigators estimate the time commitment for each round of CPV administration to be approximately 45 - 60 minutes. All responses to the cases will be completed online and will be kept confidential. Over 2 CPV administration rounds, the total time to care for the simulated patients is estimated at 1.5-2 hours.

If physicians are randomized to the intervention group in this study, they will receive educational materials on a novel diagnostic test after the first round of CPV administration. They are asked to review these materials before moving to the next CPV administration round. The time to review educational materials is estimated to be approximately 15 minutes.

Depending on the results of this randomized controlled trial, there may be an opportunity for physicians to re-enroll in a follow-on study. If they choose to participate in this second study, they will be asked to identify and send de-identified records of patients in their practice that are similar to the simulated patients they previously cared for in this study.

ELIGIBILITY:
Inclusion Criteria:

* Licensed primary care provider (PCP) (MD, DO, NP, PA) currently practicing in the following areas: a) Internal medicine b) Family medicine
* Have practiced as a PCP in internal or family medicine for greater than 2 but less than 30 years
* practicing in a community / non-academic based practice setting
* ≥ 40 patients under care weekly
* Commonly treats patients with congestive heart failure/atrial fibrillation, diabetes, hypertension, and COPD
* Practicing in the United States
* English-speaking
* Access to the internet
* Informed and voluntarily consented to be in the study

Exclusion Criteria:

* Non-English speaking
* Not a licensed primary care provider
* Unable to access the internet
* Not practicing in the U.S.
* Do not voluntarily consent to be in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Clinical Performance and Value (CPV) -measured variation in assessment | [4 months]
  Using the responses to the simulated patient cases to measure the baseline levels of variation in the work-up, recognition, and management of medication non-adherence and/or DDI in patients with more than one cardiometabolic condition and associated polypharmacy. Work-up, recognition, and management scores will be combined to report variation in total assessment of the simulated patient cases.
CPV-measured change in treatment Quality | [4 months]
  Measuring the difference in the quality of overall diagnostic scores between control participants using standard-of-care diagnostic tools and intervention participants using the CDMT. Scores will be on a scale of 0-100 with 100 representing the ideal management of a simulated patient.
CPV-measured difference in amount of evidence-based decisions | [4 months]
  Differences in number of evidence-based decisions, particularly prescribing decisions, made by intervention providers and control providers, while controlling for provider and practice characteristics, between rounds 1 and 2.

SECONDARY OUTCOMES:
CPV-measured differences in cost of care between control and intervention arms | [4 months]
  Difference in the cost of care between control and intervention participants (Cost will be calculated by measuring differential rates of medical interventions/levels of care selected by each arm, and multiplying by Medicare reimbursement rates for these interventions, and/or by modeling the incidence of expected complications and calculating associated costs per above).

CONTACTS AND LOCATIONS:
Locations (1):
- QURE Healthcare, San Francisco, California, United States